CLINICAL TRIAL: NCT07359677
Title: Effectiveness and Safety of Transcutaneous Electrical Stimulation With 40 kHz Alternating Currents in People With Spinal Cord Injury and Neuropathic Pain. A Randomised, Double-blind, Parallel Pilot Study With Placebo Control
Brief Title: High-frequency Alternating Current Stimulation for Neurophatic Pain in Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCI-Neuromodest-gifto
Record Dates: First submitted 2025-11-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain; Spinal Cord Injuries (SCI)
Keywords: High-frequency alternating current stimulation; Spinal cord injury; Neuropathic pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Two interventions will be performed:
  * Intervention A: active stimulation (High-frequency current stimulation 40kHz).
  * Intervention B: sham stimulation (simulated electrical stimulation).
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants will be performed using the same equipment, electrodes, and placement for the real or sham stimulation treatments. In addition, both the participants and the outcome assessor will not have a view of the equipment screen.
  Blinding of the outcome assessor will be performed using different team members for randomization of the interventions (Researcher 1), intervention (Researcher 2), evaluation (Researcher 3), and statistical analysis (Researcher 4). Randomization will be kept hidden from participants and research team members and only the researcher who will deliver the intervention (Researcher 2) will know the group assignment. Successful blinding of participants and evaluator will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 40 kHz (Experimental): Alternating current stimulation with a 40kHz frequency with a transcutaneous approach, 20 minutes for each intervention.
  Interventions: Device: Active group 40 kHz
- Sham stimulation (Sham Comparator): Sham stimulation via transcutaneous approach will be delivered only for the first 30 seconds, following the same procedures as the 40kHz group.
  Interventions: Device: Sham intervention

INTERVENTIONS:
Device: Active group 40 kHz — For experimental electrical stimulation, two stainless steel electrodes with conductive gel will be applied over the bilateral spinal roots with a separation between electrodes of at least 2 cm and a distance between the medial edge of each electrode and the spinous process of at least 1 cm. The upper third of the electrode will be placed above the level of spinal cord injury where the participant will have preserved sensitivity, and the remaining two thirds in the lesion and/or infralesional area. An unmodulated rectangular alternating or biphasic electrical current with a frequency of 40 kHz will be applied. The intensity of the current will be adjusted individually, increasing it until the participant reports a sensation of 'strong but comfortable tingling' just below the motor threshold. Every two minutes, the intensity of the current will be adjusted if the tingling sensation decreases. The electrical current will be applied for 20 minutes in two 10-minute phases.
  Arms: Experimental: 40 kHz
Device: Sham intervention — Placebo stimulation will be performed using the same electrical current device, the same electrode placement, and the same stimulation parameters as in the experimental stimulation, but the current intensity will be increased only during the initial 30 initial seconds and the final 30 seconds of the session, with the current intensity set to 0 mA for the rest of the intervention (20 minutes).
  Arms: Sham stimulation

SUMMARY:
To investigate the safety and effectiveness of transcutaneous electrical stimulation with 40 kHz alternating currents combined with standard treatment compared to placebo electrical stimulation plus standard treatment for neuropathic pain in people with spinal cord injury.

DETAILED DESCRIPTION:
Neuropathic pain affects more than a third of people with spinal cord injuries, reducing their quality of life, and the effectiveness of current treatments is limited. The latest research on healthy volunteers has shown that transcutaneous electrical stimulation with high-frequency blocking currents could have a potential effect on pain, proving to be a safe intervention.

To investigate the safety and effectiveness of transcutaneous electrical stimulation with 40 kHz alternating currents combined with standard treatment compared to placebo electrical stimulation plus standard treatment for neuropathic pain in people with spinal cord injury.

Design: Parallel, randomised, double-blind, placebo-controlled pilot clinical trial.

Participants and location: People with spinal cord injury over the age of 18, with a history of more than three months, neuropathic pain at the level of injury and/or below the level of injury, and pain intensity ≥ 30 mm on the visual analogue scale (VAS) for pain. Participants with any contraindications for the application of transcutaneous electrical stimulation will be excluded. The study will be conducted at the National Hospital for Paraplegics in Toledo.

Intervention: Participants will be randomly assigned to two intervention groups:

Active group (n=15) transcutaneous electrical stimulation with 40kHz alternating currents and Placebo group (n=15) simulated stimulation. The duration of the session in both interventions will be 20 minutes, 10 sessions, over two weeks (5 sessions/week).

Main variables and measurement instruments: The main variable will be the Spanish version of the Neuropathic Pain Symptom Inventory. Secondary variables will be pain perception, which will be assessed using a daily record of spontaneous pain with the VAS scale. The intensity of pain evoked by mechanical stimuli will be assessed using the VAS scale, and pain evoked by thermal stimuli will be assessed using a quantitative sensory test with a Peltier thermode. An ad hoc questionnaire has been designed to assess adverse effects. The assessments will be carried out at four time points: before the intervention, during the intervention, immediately after the intervention, and one week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* People with spinal cord injuries of any aetiology affecting the D1 spinal cord level or lower (paraplegia)
* With injury grade A, B, C, or D according to the ASIA (American Spinal Injury Association) Impairment Scale (AIS)
* Time since spinal cord injury ≥ 3 months
* A score of ≥ 4 points on the Dolour Neuropathique 4 (DN4) scale
* Neuropathic pain at the level of the injury (within the dermatome at that level and up to three dermatomes below) and/or below the level of the injury (more than three dermatomes below)
* Duration of pain ≥ 1 month
* Average pain perception score ≥ 30 mm on the visual analogue scale (VAS) in the week prior to eligibility, with a daily record of 5 days (Monday to Friday) in the morning.
* Be able to understand instructions and assessment tools
* Agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Cauda equina injuries
* Brain injuries or other central nervous system injuries concomitant with spinal cord injury
* A value of 100 mm in any of the daily records collected in the week prior to eligibility
* Having any contraindications for the application of transcutaneous electrical stimulation: cardiac pacemaker or any other implanted electrical device, epilepsy, pregnancy, active malignant tumours in the area of application of the stimulation, and wounds or skin damage in the area of stimulation
* History of psychiatric illness
* Major depression
* Spinal cord injury caused by autolysis
* Changes in medication prescribed for the treatment of pain and spasticity during the study
* Acute nociceptive pain in any area of the body during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain perception - NPSI | Prior to the intervention (Baseline), during the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  It will be assessed using the Spanish version of the Neuropathic Pain Symptom Inventory (NPSI), and the result will be taken as the change from baseline at different time points.
  This questionnaire has a score ranging from 0 to 100 points, with a higher score indicating greater severity of neuropathic pain symptoms. Regarding the psychometric properties of this questionnaire, it has been shown that the areas under the receiver operating characteristic curves were greater than 0.85 and all reliability coefficients were greater than 0.70.

SECONDARY OUTCOMES:
Pain perception - VAS | Baseline (-5 to 0 days), week 1 treatment (days 1-5), week 2 treatment (days 6-10) and post-treatment week (days 11-15).
  A daily assessment (Monday to Friday) will be carried out in the morning of self-perceived pain using the visual analogue scale (VAS) (0 mm no pain and 100 mm maximum imaginable pain). The result will be taken as the change from baseline in the weekly mean value of self-perceived pain.
Change in pain threshold evoked by mechanical stimuli | Prior to the intervention (Baseline), during the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  The change in pain threshold evoked by mechanical stimuli will be assessed at and below the level of injury-specifically, within the dermatome of the lesion and up to three dermatomes below, and in areas more than three dermatomes below the lesion. Mechanical allodynia will be evaluated using the SenseLab™ Brush-05 (Somedic, Sweden), with two 40 mm brush strokes applied 2 seconds apart. Pinprick pain will be assessed using three stimuli with a 512 mN Von Frey filament no. 12 (OptiHair 2, Germany). In both cases, pain intensity will be rated using a 0-100 mm Visual Analogue Scale (VAS).
Change in pain threshold evoked by thermal (cold and heat) stimuli | Prior to the intervention (Baseline), during the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  The change in pain threshold evoked by thermal (cold and heat) stimuli will be assessed at and below the level of injury-specifically, within the dermatome of the lesion and up to three dermatomes below, and in areas more than three dermatomes below the lesion. Thermal pain thresholds will be measured using a 32 × 32 mm Peltier thermode (TSA 2, MEDOC, Israel), with temperature changes from a 30 °C baseline at 1 °C/s. Heat and cold pain thresholds will be recorded using the method of limits, taking the average of three consecutive stimuli. For safety, maximum and minimum cut-offs will be set at 50 °C and 0 °C, respectively.
Patient's Overall Impression of Change | During the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  A record of the Global Patient Change Rating Scale will be made at post-treatment and during follow-up with respect to the baseline situation. This scale consists of 7 items ranging from '1 = much better' to '7 = much worse'.
Percentage of participants responding to treatment | Baseline (-5 to 0 days), week 1 treatment (days 1-5), week 2 treatment (days 6-10) and post-treatment week (days 11-15).
  The percentage of participants responding to treatment will be evaluated as those who achieve a reduction in pain in the weekly Visual Analog Scale average ≥ 30% and ≥ 50% after treatment and at follow-up.
Pain interference with sleep | Baseline (-5 to 0 days), week 1 treatment (days 1-5), week 2 treatment (days 6-10) and post-treatment week (days 11-15).
  Pain interference with sleep will be reported in a daily morning log (Monday to Friday) using the VAS scale (0 mm = pain does not interfere with sleep and 100 mm = pain completely interferes with sleep) The result will be taken as the change from baseline in the weekly mean value of pain interference with sleep.
Spasticity | Prior to the intervention (Baseline), during the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  To this end, the Modified Ashworth Scale will be used to assess resistance to passive movement in the knee joint bilaterally. The Modified Ashworth Scale ranges from a minimum score of 0 to a maximum score of 4 and is used to assess the degree of muscle spasticity. Higher scores indicate worse outcomes.
Frequency of spasms | Prior to the intervention (Baseline), during the intervention after five sessions (Day 5), after the intervention (Day 10) and one week after the end of the intervention (Day 15)
  The Penn Spasm Frequency Scale ranges from a minimum score of 0 to a maximum score of 4 and evaluates the frequency of muscle spasms. Higher scores indicate worse outcomes, reflecting more frequent and severe spasms.
Adverse events | Week 1 treatment (days 1-5), week 2 treatment (days 6-10)
  Adverse effects related to the electrical current will be recorded using an ad hoc questionnaire specifically designed for this study.

OTHER OUTCOMES:
Success of blinding | Day 10
  The success of blinding the participants and evaluators will be assessed using a question with five response options: "What type of intervention do you think you have received?": "I strongly believe that I received an experimental treatment
  / I slightly believe that I received an experimental treatment / I strongly believe that I received a placebo / I slightly believe that I received a placebo / I don't know / No answer

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Principal Investigator — Castilla La Mancha University
Locations (1):
- Hospital Nacional de Parapléjicos, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No